CLINICAL TRIAL: NCT05955079
Title: Prospective Validation of the Association Between Circulating Tumor DNA Detection and Risk of Metastatic Relapse in Patients With Localized Endometrial Cancer
Brief Title: Circulating Tumor DNA Study in Patients With Endometrial Cancer
Acronym: ctDNA-endo
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: CARPEM, Institut du Cancer Paris (Unknown); Centre de recherche des Cordeliers (Unknown); METHYS DX (Unknown)
Responsible Party: Sponsor
Other Study IDs: CRC22003; 20200812151455 (Other: AP-HP)
Record Dates: First submitted 2023-07-12; First posted 2023-07-21 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-05

CONDITIONS: Endometrial Cancer
Keywords: Endometrial Cancer; Digital-PCR; Circulating Tumor DNA; minimal residual disease; liquid biopsy
MeSH Terms: conditions — Endometrial Neoplasms; Neoplasm, Residual

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, three samples (before, after surgery and before chemotherapy)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Endometrial Cancer: Patients over 18 years old with a biopsy-proven endometrial cancer, at FIGO stage I to IV, and amenable and undergoing surgical treatment
  Interventions: Other: Whole blood

INTERVENTIONS:
Other: Whole blood — 3 samples (before, after surgery and before chemotherapy)

SUMMARY:
The objective of this study is to identify a population at risk of early recurrence after oncologic resection surgery of a primary uterine tumor based on the detection of ctDNA

DETAILED DESCRIPTION:
Despite early management, the risk of recurrence in non-metastatic endometrial cancer (FIGO I-III) is approximately 10-20%. The challenge is to identify the most high-risk cases for relapse in order to adapt surgical and medical management.

The development of digital PCR methods in nano-droplets, detecting circulating tumor DNA (ctDNA) with high sensitivity, could help to better specify the prognosis of patients with localized endometrial cancer and to identify a population with residual disease, the source of this ctDNA.

The investigators established a universal methylation signature in the laboratory based on analysis of endometrial cancer-specific DNA methylation using in silico analysis of public data from the Cancer Genome Atlas, validated in an independent cohort, with 99% sensitivity and 98% specificity.

A prospective biological cohort was established between the gynecology and medical oncology departments and the Cochin Hospital biological resources center (CARPEM-OncoCentre collection).

This is a prospective monocentric biological collection study.

The aim of this study is to evaluate the prognostic impact of pre- and post-operative ctDNA detection in stage I-III endometrial cancer.

ELIGIBILITY:
Inclusion Criteria:

* Female patients over 18 years of age who are potentially eligible for inclusion in the OncoCentre collection (registered as a patient at APHP, without legal protection measures, affiliated with a social security system)
* Patients diagnosed with histologically documented endometrial cancer on an endometrial biopsy
* Surgical intervention performed at Hopital Cochin

Exclusion Criteria:

* Failure to sign the OncoCentre consent form
* Refusal of OncoCentre consent
* Patient not eligible for upfront curative surgical treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women undergoing clinically-indicated hysterectomy for endometrial cancer at the University Paris Cité hospital Cochin, who are age 18 years and older
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Recurrence-free survival | 1 year

SECONDARY OUTCOMES:
Recurrence-free survival | 3 years
Frequency of ctDNA detection based on established prognostic parameters | 3 years
  Frequency of ctDNA detection based on established prognostic parameters: histological type (endometrioid, non-endometrioid), grade (low grade, high grade), stage (localized to the uterus stages I-II or stage III with nodal involvement), lymphovascular invasion (present/absent), and molecular group (low risk: POLE, intermediate risk: MSI/NSMP, high risk: TP53).
Frequency of ctDNA detection in other prognostic groups | 3 years
  Frequency of ctDNA detection in other prognostic groups according to the 2021 ESGO-ESTRO-ESP classification
Frequency of ctDNA detection based on the recurrence profile | 3 years
  Frequency of ctDNA detection based on the recurrence profile : anatomical (locoregional versus distant; abdominal versus extra-abdominal; visceral or nodal) or dynamic (aggressive recurrence (progression-free survival post recurrence <6 months) or non-aggressive (>6 months))

CONTACTS AND LOCATIONS:
Overall Officials: Bruno BORGHESE, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris; Jérôme ALEXANDRE, MD, PhD, Study Chair — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Cochin, Paris, France

REFERENCES:
- [Background] Beinse G, Borghese B, Metairie M, Just PA, Poulet G, Garinet S, Parfait B, Didelot A, Bourreau C, Agueeff N, Lavolle A, Terris B, Chapron C, Goldwasser F, Leroy K, Blons H, Laurent-Puig P, Taly V, Alexandre J. Highly Specific Droplet-Digital PCR Detection of Universally Methylated Circulating Tumor DNA in Endometrial Carcinoma. Clin Chem. 2022 Jun 1;68(6):782-793. doi: 10.1093/clinchem/hvac020. PMID 35323926
- [Background] Lu KH, Broaddus RR. Endometrial Cancer. N Engl J Med. 2020 Nov 19;383(21):2053-2064. doi: 10.1056/NEJMra1514010. No abstract available. PMID 33207095
- [Background] Morice P, Leary A, Creutzberg C, Abu-Rustum N, Darai E. Endometrial cancer. Lancet. 2016 Mar 12;387(10023):1094-1108. doi: 10.1016/S0140-6736(15)00130-0. Epub 2015 Sep 6. PMID 26354523
- [Background] Cancer Genome Atlas Research Network; Kandoth C, Schultz N, Cherniack AD, Akbani R, Liu Y, Shen H, Robertson AG, Pashtan I, Shen R, Benz CC, Yau C, Laird PW, Ding L, Zhang W, Mills GB, Kucherlapati R, Mardis ER, Levine DA. Integrated genomic characterization of endometrial carcinoma. Nature. 2013 May 2;497(7447):67-73. doi: 10.1038/nature12113. PMID 23636398
- [Background] Leon-Castillo A, de Boer SM, Powell ME, Mileshkin LR, Mackay HJ, Leary A, Nijman HW, Singh N, Pollock PM, Bessette P, Fyles A, Haie-Meder C, Smit VTHBM, Edmondson RJ, Putter H, Kitchener HC, Crosbie EJ, de Bruyn M, Nout RA, Horeweg N, Creutzberg CL, Bosse T; TransPORTEC consortium. Molecular Classification of the PORTEC-3 Trial for High-Risk Endometrial Cancer: Impact on Prognosis and Benefit From Adjuvant Therapy. J Clin Oncol. 2020 Oct 10;38(29):3388-3397. doi: 10.1200/JCO.20.00549. Epub 2020 Aug 4. PMID 32749941
- [Background] Kommoss S, McConechy MK, Kommoss F, Leung S, Bunz A, Magrill J, Britton H, Kommoss F, Grevenkamp F, Karnezis A, Yang W, Lum A, Kramer B, Taran F, Staebler A, Lax S, Brucker SY, Huntsman DG, Gilks CB, McAlpine JN, Talhouk A. Final validation of the ProMisE molecular classifier for endometrial carcinoma in a large population-based case series. Ann Oncol. 2018 May 1;29(5):1180-1188. doi: 10.1093/annonc/mdy058. PMID 29432521
- [Background] Colombo N, Creutzberg C, Amant F, Bosse T, Gonzalez-Martin A, Ledermann J, Marth C, Nout R, Querleu D, Mirza MR, Sessa C; ESMO-ESGO-ESTRO Endometrial Consensus Conference Working Group. ESMO-ESGO-ESTRO Consensus Conference on Endometrial Cancer: diagnosis, treatment and follow-up. Ann Oncol. 2016 Jan;27(1):16-41. doi: 10.1093/annonc/mdv484. Epub 2015 Dec 2. PMID 26634381
- [Background] de Boer SM, Powell ME, Mileshkin L, Katsaros D, Bessette P, Haie-Meder C, Ottevanger PB, Ledermann JA, Khaw P, Colombo A, Fyles A, Baron MH, Jurgenliemk-Schulz IM, Kitchener HC, Nijman HW, Wilson G, Brooks S, Carinelli S, Provencher D, Hanzen C, Lutgens LCHW, Smit VTHBM, Singh N, Do V, D'Amico R, Nout RA, Feeney A, Verhoeven-Adema KW, Putter H, Creutzberg CL; PORTEC study group. Adjuvant chemoradiotherapy versus radiotherapy alone for women with high-risk endometrial cancer (PORTEC-3): final results of an international, open-label, multicentre, randomised, phase 3 trial. Lancet Oncol. 2018 Mar;19(3):295-309. doi: 10.1016/S1470-2045(18)30079-2. Epub 2018 Feb 12. PMID 29449189
- [Background] Corcoran RB, Chabner BA. Application of Cell-free DNA Analysis to Cancer Treatment. N Engl J Med. 2018 Nov 1;379(18):1754-1765. doi: 10.1056/NEJMra1706174. No abstract available. PMID 30380390
- [Background] Phallen J, Sausen M, Adleff V, Leal A, Hruban C, White J, Anagnostou V, Fiksel J, Cristiano S, Papp E, Speir S, Reinert T, Orntoft MW, Woodward BD, Murphy D, Parpart-Li S, Riley D, Nesselbush M, Sengamalay N, Georgiadis A, Li QK, Madsen MR, Mortensen FV, Huiskens J, Punt C, van Grieken N, Fijneman R, Meijer G, Husain H, Scharpf RB, Diaz LA Jr, Jones S, Angiuoli S, Orntoft T, Nielsen HJ, Andersen CL, Velculescu VE. Direct detection of early-stage cancers using circulating tumor DNA. Sci Transl Med. 2017 Aug 16;9(403):eaan2415. doi: 10.1126/scitranslmed.aan2415. PMID 28814544
- [Background] Bolivar AM, Luthra R, Mehrotra M, Chen W, Barkoh BA, Hu P, Zhang W, Broaddus RR. Targeted next-generation sequencing of endometrial cancer and matched circulating tumor DNA: identification of plasma-based, tumor-associated mutations in early stage patients. Mod Pathol. 2019 Mar;32(3):405-414. doi: 10.1038/s41379-018-0158-8. Epub 2018 Oct 12. PMID 30315273
- [Background] Shintani D, Hihara T, Ogasawara A, Sato S, Yabuno A, Tai K, Fujiwara K, Watanabe K, Hasegawa K. Tumor-related mutations in cell-free DNA in pre-operative plasma as a prognostic indicator of recurrence in endometrial cancer. Int J Gynecol Cancer. 2020 Sep;30(9):1340-1346. doi: 10.1136/ijgc-2019-001053. Epub 2020 Jul 21. PMID 32699017
- [Background] Taieb J, Taly V, Henriques J, Bourreau C, Mineur L, Bennouna J, Desrame J, Louvet C, Lepere C, Mabro M, Egreteau J, Bouche O, Mulot C, Hormigos K, Chaba K, Mazard T, de Gramont A, Vernerey D, Andre T, Laurent-Puig P. Prognostic Value and Relation with Adjuvant Treatment Duration of ctDNA in Stage III Colon Cancer: a Post Hoc Analysis of the PRODIGE-GERCOR IDEA-France Trial. Clin Cancer Res. 2021 Oct 15;27(20):5638-5646. doi: 10.1158/1078-0432.CCR-21-0271. Epub 2021 Jun 3. PMID 34083233
- [Background] Shen H, Laird PW. Interplay between the cancer genome and epigenome. Cell. 2013 Mar 28;153(1):38-55. doi: 10.1016/j.cell.2013.03.008. PMID 23540689
- [Background] Garrigou S, Perkins G, Garlan F, Normand C, Didelot A, Le Corre D, Peyvandi S, Mulot C, Niarra R, Aucouturier P, Chatellier G, Nizard P, Perez-Toralla K, Zonta E, Charpy C, Pujals A, Barau C, Bouche O, Emile JF, Pezet D, Bibeau F, Hutchison JB, Link DR, Zaanan A, Laurent-Puig P, Sobhani I, Taly V. A Study of Hypermethylated Circulating Tumor DNA as a Universal Colorectal Cancer Biomarker. Clin Chem. 2016 Aug;62(8):1129-39. doi: 10.1373/clinchem.2015.253609. Epub 2016 Jun 1. PMID 27251038
- [Background] Kint S, De Spiegelaere W, De Kesel J, Vandekerckhove L, Van Criekinge W. Evaluation of bisulfite kits for DNA methylation profiling in terms of DNA fragmentation and DNA recovery using digital PCR. PLoS One. 2018 Jun 14;13(6):e0199091. doi: 10.1371/journal.pone.0199091. eCollection 2018. PMID 29902267
- See also: Related Info — https://carpem.fr/activites/les-plateformes/biobanques/projets-de-recherche-collection-oncocentre/